CLINICAL TRIAL: NCT00682682
Title: Reducing Brief Thermal and Electrical Pain (Four Study Days)
Acronym: 4DO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Chris Hoffer, Research Coordinator, University of Washington
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 030091D
Record Dates: First submitted 2008-05-20; First posted 2008-05-22 (Estimated); Last update posted 2011-09-13 (Estimated); Status verified 2011-09

CONDITIONS: Pain
Keywords: Pain distraction; Analgesic interventions; Burn patients
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): all study participants will have 4 visits: VR alone, VR + opioid, opioid alone, and no VR/opioid
  Interventions: Other: Virtual Reality video distraction; Other: Virtual Reality video game

INTERVENTIONS:
Other: Virtual Reality video distraction — Virtual Reality involves wearing a helmet and playing a game called "Snow world". This game has sound and is presented in 3D format. This game has immersive qualities that help user feel as if they are "in" the game.
Other: Virtual Reality video game — Virtual Reality video games involve wearing a helmet with vision and sound. this game is presented in 3D which gives the user the feeling of being "in" the game. The game used for this study is "Snow World"

SUMMARY:
Ultimately, the purpose of the present study is to help improve pain control in burn patients during wound care and physical therapy, where pain levels with opioids alone are often excessively high.

This study measures how much virtual reality pain distraction reduces pain compared to traditional opioid pain meds, and whether there is additional pain reduction when Virtual Reality distraction + Opioids are combined. In addition to studying the amount of pain reduction, this study will also measure side effects (if any) of the two treatments (Virtual Reality pain distraction and Opioids) alone and when combined.

Healthy volunteers will be recruited from advertisements will undergo a trial of the pain testing. They will receive a series of brief stimuli (at a painful but tolerable safe intensities they select and approve during baseline testing), separated by intervals of no pain.

Participants will rate how much pain they felt after each brief stimulus, and will fill out side effects questionnaires after finishing the pain session.

Subjects will participate in each of the four conditions in which the order is randomized.

* No opioids (0ng/ml hydromorphone) + no virtual reality Snow World distraction
* No opioids + yes virtual reality Snow World distraction
* Moderate dose of pain medicine (4ng/ml hydromorphone) + no virtual reality
* Moderate dose of pain medicine + yes virtual reality Snow World distraction

It is our hypothesis that VR distraction + opioids will show a reduced perception of pain in subjects more than opioids alone or no intervention (control).

DETAILED DESCRIPTION:
In this study, healthy volunteers aged 18-45 who sign up after seeing a flyer or web posting are screened for exclusion via telephone interview, and if eligible, a health background interview. Initial contact will come from the subject's response to recruitment materials. Subjects may withdraw at any time.

These safe laboratory studies with healthy volunteers are designed to help us figure out how to maximize the effectiveness of virtual reality when used with severe burn patients at Harborview Burn Center

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women 18-45 years old
* Normal height and weight ratio

Exclusion Criteria:

* women who are pregnant and nursing
* history of substance abuse
* access to opioids in the workplace
* smokes cigarettes
* history of medical problems with the following: heart, lungs, liver, kidneys, endocrine, neurologic, migraines, or psychiatric requiring medical intervention
* anemia
* chronic pain
* allergy or hypersensitivity to opioids, velcro, or latex
* severe motion sickness
* unusual sensitivity or lack of sensitivity to pain
* sensitive skin or feet

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2007-12; Primary Completion 2008-05 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Efficacy of VR distraction with and without opioid when pain stimulus is applied. | at completion of study

CONTACTS AND LOCATIONS:
Overall Officials: Samuel R. Sharar, MD, Principal Investigator — Professor, University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States